CLINICAL TRIAL: NCT02392468
Title: Randomised, Parallel-group, Double-blind Study of Systemic and Ocular Safety and Pharmacokinetics of BI 409306 in Patients With Schizophrenia, Alzheimer's Disease, and Age-comparable Healthy Volunteers
Brief Title: Study of Systemic and Ocular Safety and Pharmacokinetics of BI 409306 in Patients With Schizophrenia, Alzheimer's Disease, and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.27
Record Dates: First submitted 2015-03-17; First posted 2015-03-19 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Alzheimer Disease
MeSH Terms: conditions — Schizophrenia; Alzheimer Disease | interventions — BI 409306

ARMS (6):
- BI 409306 25 milligram (mg) - Alzheimer patients (Experimental): Alzheimer patients received once daily (QD) orally one tablet of 25 mg of BI 409306 and two 50 mg matching placebo tablets for 14 days.
  Interventions: Drug: Placebo matching BI 409306 50 mg; Drug: BI 409306 25 mg
- BI 409306 100 mg - Alzheimer patients (Experimental): Alzheimer patients received once daily (QD) orally 100 mg of BI 409306 (two 50 mg active tablets) and one 25 mg matching placebo tablet for 14 days.
  Interventions: Drug: Placebo matching BI 409306 25 mg; Drug: BI 409306 50 mg
- BI 409306 25 mg - Schizophrenia patients (Experimental): Schizophrenia patients (cognitive impairment associated with schizophrenia) received once daily (QD) orally one tablet of 25 mg of BI 409306 and two 50 mg matching placebo tablets for 14 days.
  Interventions: Drug: Placebo matching BI 409306 50 mg; Drug: BI 409306 25 mg
- BI 409306 100 mg - Schizophrenia patients (Experimental): Schizophrenia patients (cognitive impairment associated with schizophrenia) received once daily (QD) orally 100 mg of BI 409306 (two 50 mg active tablets) and one 25 mg matching placebo tablet for 14 days.
  Interventions: Drug: Placebo matching BI 409306 25 mg; Drug: BI 409306 50 mg
- BI 409306 25 mg - Healthy volunteers (Active Comparator): Age-comparable healthy volunteers received once daily (QD) orally one tablet of 25 mg of BI 409306 and two 50 mg matching placebo tablets for 14 days.
  Interventions: Drug: Placebo matching BI 409306 50 mg; Drug: BI 409306 25 mg
- BI 409306 100 mg - Healthy volunteers (Active Comparator): Age-comparable healthy volunteers received once daily (QD) 100 mg of BI 409306 (two 50 mg active tablets) and one 25 mg matching placebo tablet orally for 14 days.
  Interventions: Drug: Placebo matching BI 409306 25 mg; Drug: BI 409306 50 mg

INTERVENTIONS:
Drug: Placebo matching BI 409306 25 mg — Film-coated tablet
  Arms: BI 409306 100 mg - Alzheimer patients; BI 409306 100 mg - Healthy volunteers; BI 409306 100 mg - Schizophrenia patients
Drug: Placebo matching BI 409306 50 mg — Film-coated tablet
  Arms: BI 409306 25 mg - Healthy volunteers; BI 409306 25 mg - Schizophrenia patients; BI 409306 25 milligram (mg) - Alzheimer patients
Drug: BI 409306 25 mg — Film-coated tablet
  Arms: BI 409306 25 mg - Healthy volunteers; BI 409306 25 mg - Schizophrenia patients; BI 409306 25 milligram (mg) - Alzheimer patients
Drug: BI 409306 50 mg — Film-coated tablet
  Arms: BI 409306 100 mg - Alzheimer patients; BI 409306 100 mg - Healthy volunteers; BI 409306 100 mg - Schizophrenia patients

SUMMARY:
Single site, parallel-group, double-blind trial of low or high dose of BI 409306 to evaluate the ocular and systemic safety and pharmacokinetics during 14 day treatment period in patients with schizophrenia, Alzheimer's disease, or age comparable healthy volunteers.

ELIGIBILITY:
Inclusion criteria:

* Schizophrenia group:

  * Patients with established diagnoses of schizophrenia (per Diagnostic and Statistic Manual of Mental Disorder, version V) with the all of the following clinical features:

    * Clinically stable and are in the residual (non-acute) phase of their illness for at least 8 weeks prior to randomisation
    * Current antipsychotic and concomitant psychotropic medications must meet the criteria below:

      * Maintained on current atypical (second generation) antipsychotic medications (in any approved dosage form) other than Clozapine and on current dose for at least 8 weeks prior to randomisation, and/or
      * Maintained on current typical (first generation) antipsychotic medications and on current dose for at least 6 months, optionally combined with anticholinergics if treated with a stable dose for at least 6 months prior to randomisation, and/or
      * Maintained on current concomitant psychotropic medications other than anticholinergics, antiepileptics and lithium, and on current dose for at least 8 weeks prior to randomisation. Antiepileptics and lithium are allowed if initiated at least 6 months prior to randomisation.
    * Have no more than a moderate severity rating on hallucinations and delusions (Positive and Negative Syndrome Scale (PANSS), positive syndrome Hallucinatory Behavior item score <= 4 and Delusions item score <= 4)
    * Have no more than a moderate severity rating on positive formal thought disorder (PANSS, positive syndrome Conceptual Disorganization item score <= 4)
    * Have a minimal level of extrapyramidal symptoms (Simpson-Angus Scale total score < 6) and depressive symptoms (PANSS, general psychopathology syndrome Depression item score <= 4)
  * Male or female patients age 18 to 55 years.
* Alzheimer's Disease group:

  * Patients with diagnosis of mild Alzheimer's Dementia based on DSM-V and in accordance with the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease.
  * Mini-Mental State Examination (MMSE) score of 18-26.
  * Male or female patients age 55 to 85 years, who have not been taking acetyl cholinesterase inhibitors (donepezil, galantamine, rivastigmine) and/or memantine for at least 3 months or on stable dose of acetyl cholinesterase inhibitors (donepezil, galantamine, rivastigmine) and/or memantine at least 3 months before randomization.Patients older than 85 years may be included based on an acceptable general health status, (e.g. concomitant diseases, physical capability to follow the required study procedures [visits etc.]) per investigators judgement.
  * Availability of a pre-existing cranial computer tomography (CCT) or magnetic resonance imaging (MRI) scan of the brain (initiation of radiological imaging is not required) not older than one year prior to screening; if not available, a CCT must be performed at screening. Results of radiological brain imaging must be compatible with Diagnosis of Alzheimer's Disease and exclusion of relevant signs indicative of potential vascular dementia (see also exclusion criteria).
  * If needed, a caregiver may be present during site activities.
* Age-comparable male or female healthy volunteers age 18 to 85 years. Healthy volunteers older than 85 years may be included based on an acceptable general health status, (e.g. concomitant diseases, physical capability to follow the required study procedures [visits etc.]) per investigators judgement:

  * After 10 patients with schizophrenia (as described above) are entered into the study, the median age of the group will be computed. Five healthy volunteers at or below the median age but greater than 18 years old and five healthy volunteers above the median but less than 55 will be entered into the study.
  * Similarly, after 10 patients with AD are entered, the median age will be computed. Five healthy volunteers at or below the median age but greater than 55 years old and five healthy volunteers above the median but less than 85 will be entered into the study.
* Subjects must exhibit reliability and physiologic capability to comply with all protocol procedures.
* Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice and the local legislation. If the patient needs a legal representative, then this legal representative must give written informed consent as well.

Exclusion criteria:

* Presence of active ocular conditions with or without visual impairment due to any causes (e.g. cataract, chorioretinal macular lesion, amblyopia, active diabetic retinopathy, uncontrolled glaucoma, active inflammation or infection, etc.) in one eye or both eyes at the screening phase.
* Planned ocular treatment (e.g. intravitreal antivascular growth factor, corticosteroids) or surgery during the study period.
* Current or planned use of ocular or systemic corticosteroids.
* Current or planned use of medications known to be toxic to the retina, lens, optic nerve
* Subjects treated with more than two antipsychotic medications (including more than two dosage forms).
* Dementia in Alzheimers Disease patients, secondary to other disorders (based on clinical data and/or current laboratory findings and/or on a pre-existing cranial MRI or CCT).
* Neurological disease (other than Dementia of Alzheimer Type such as: Lewy body dementia - primary diagnosis, Huntington's disease, Parkinson's Disease encephalitis, epilepsy, vascular or multi-infarct dementia, stroke, congenital mental deficiency, or multiple sclerosis), or mental retardation.
* Subjects needing to take long-acting hypnotics or anxiolytic (i.e. Diazepam).
* For AD patients, the following drugs are prohibited for 3 months prior to randomization and for the duration of the trial:

  * tricyclic antidepressants,
  * antidepressants that are monoamine oxidase inhibitors,
  * neuroleptics with moderate or greater anticholinergic potency (e.g., chlorpromazine, fluphenazine, loxapine, perphenazine, thioridazine),
  * anticholinergic medications.
  * Intake of St. John's wort, Carbamazepine and extracts from Ginko as they are relevant CYP2C19 inducers.
* Substantial concomitant cerebrovascular disease (defined by a history of a stroke/intracranial haemorrhagia temporally related to the onset of worsening of cognitive impairment).
* Any suicidal ideation of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS) in the past 3 months.
* Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
* History or diagnosis of symptomatic and unstable/uncontrolled gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, haematological or hormonal disorders.
* For female subjects:

  --Pre-menopausal women (last menstruation <=1 year prior to informed consent) who:
  * are nursing or pregnant or
  * are of child-bearing potential and are not practicing an acceptable method of birth control
* For male subjects: Men who are able to father a child, unwilling to be abstinent or use adequate contraception.
* Known history, or new diagnosis of HIV infection.
* Significant renal disease (CLCR < 30 mL/min).
* Bodyweight < 50 kg.
* Indication of liver disease.
* History of neurologic (e.g. stroke, seizure without a clear and resolved etiology, concussion accompanying loss of consciousness) or psychiatric condition.
* History of malignancy within the last 5 years, except for basal cell carcinoma.
* Planned elective surgery requiring general anaesthesia, or hospitalisation during the study period.
* Significant history of drug dependence
* Clinically significant uncompensated hearing loss. Use of hearing aids is not allowed.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- United States (3):
  - University of California San Diego, La Jolla, California
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Community Clinical Research, Inc., Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The randomised, parallel-group, double-blind study of systemic and ocular safety and pharmacokinetics of BI 409306 in patients with schizophrenia, Alzheimer's disease, and age-comparable healthy volunteers
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
Started | 10 | 11 | 10 | 10 | 9 | 11
Completed | 10 | 10 | 10 | 10 | 9 | 10
Not Completed | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all participants who were documented to have been administered at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers | Total
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 9 | 11 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 74.5 (9.2) | 77.8 (8.6) | 40.5 (9.1) | 35.1 (7.8) | 55.9 (22.4) | 60.2 (21.6) | 57.7 (21.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 6 | 8 | 2 | 2 | 4 | 5 | 27
    Male | 4 | 3 | 8 | 8 | 5 | 6 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Hispanic or Latino | 0 | 2 | 1 | 1 | 4 | 2 | 10
    Not Hispanic or Latino | 10 | 9 | 9 | 9 | 5 | 9 | 51
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 1 | 0 | 0 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 6 | 5 | 2 | 2 | 15
    White | 9 | 11 | 3 | 5 | 7 | 9 | 44
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Adverse Events (AEs), Coded to the Medical Dictionary for Regulatory Activities - System Organ Class Eye Disorders, as Determined by the Investigator at the End of Trial
Description: The percentage of participants with Adverse Events (AEs), coded to the Medical Dictionary for Regulatory Activities (MedDRA) - System Organ Class (SOC) 'Eye disorders', as determined by the investigator at the End of Trial (EOT) is reported.
  Percentages were rounded to one decimal place.
Time Frame: From the first dose of trial medication until 7 days after last in-take of trial medication, 21 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 9 | 11
Percentage of participants | 40.0 | 27.3 | 0.0 | 20.0 | 22.2 | 72.7

2. Secondary Outcome: The Percentage of Participants With Drug-related AEs as Determined by the Investigator at EOT
Description: The percentage of participants with drug-related adverse events (AEs) as determined by the investigator at end of trial (EOT) is reported.
  Percentages were rounded to one decimal place.
Time Frame: From the first dose of trial medication until 7 days after last in-take of trial medication, 21 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 9 | 11
Percentage of participants | 30.0 | 36.4 | 0.0 | 20.0 | 33.3 | 81.8

3. Secondary Outcome: Maximum Measured Concentration of BI 409306 in Plasma at Steady-state (Cmax,ss)
Description: Maximum measured concentration of BI 409306 in plasma at steady-state (Cmax,ss) is reported.
Time Frame: Pharmacokinetic blood samples were taken at 2:00 (hours: minutes) before and 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 4:00, 6:00 (hours: minutes) after drug administration on day 14.
Population: The Pharmacokinetic (PK) set (PKS) included all participants in the TS who provided at least 1 evaluable observation for at least 1 PK endpoint without important protocol violations relevant to the evaluation of PK. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per litre (nmol/L)
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
nanomoles per litre (nmol/L) | 696 (86.6) | 2290 (115.0) | 202 (72.1) | 1050 (60.4) | 466 (37.5) | 1550 (153.0)

4. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 409306 in Plasma at Steady-state (Tmax,ss)
Description: Time from dosing to maximum measured concentration of BI 409306 in plasma at steady-state (tmax,ss) is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Hours | 0.750 [0.500 to 2.000] | 1.000 [0.333 to 4.000] | 0.500 [0.333 to 1.500] | 0.525 [0.333 to 1.500] | 0.500 [0.333 to 4.000] | 0.917 [0.333 to 4.000]

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication until 7 days after last in-take of trial medication, 21 days.
Description: The residual effect period (REP) was defined as 7 days after the last trial medication intake. All adverse events which occurred through the treatment phase and throughout the REP were considered as on treatment.
  The treated set (TS) included all participants who were documented to have been administered at least 1 dose of investigational treatment.
Arm/Group | BI 409306 25 Milligram (mg) - Alzheimer Patients | BI 409306 100 mg - Alzheimer Patients | BI 409306 25 mg - Schizophrenia Patients | BI 409306 100 mg - Schizophrenia Patients | BI 409306 25 mg - Healthy Volunteers | BI 409306 100 mg - Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 6/10 | 6/11 | 6/10 | 4/10 | 5/9 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 25 Milligram (mg) - Alzheimer Patients (N=10) | BI 409306 100 mg - Alzheimer Patients (N=11) | BI 409306 25 mg - Schizophrenia Patients (N=10) | BI 409306 100 mg - Schizophrenia Patients (N=10) | BI 409306 25 mg - Healthy Volunteers (N=9) | BI 409306 100 mg - Healthy Volunteers (N=11)
Chromatopsia (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 4
Cyanopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 3
Visual brightness (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 3
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 2
Xanthopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 2 | 1 | 2 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chloropsia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02392468/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02392468/SAP_001.pdf